CLINICAL TRIAL: NCT00986713
Title: Value of Amphotericin B Inhalation for Prophylaxis of Invasive Pulmonary Aspergillosis After Renal Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Bin Cao,doctor, Beijing Chaoyang Hospital,Affiliate of Capital Medical Unibersity
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CYH-CMU AmB Neph
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Invasive Pulmonary Aspergillosis
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis | interventions — Amphotericin B

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Amphotericin B — Aerosolized Amphotericin B,2mg/day or 10mg/day

SUMMARY:
The purpose of this study is to determine whether inhalation with aerosolized amphoterin B 10mg/d is more effective than aerosolized amphoterin B 2mg/d to reduce the incidence of invasive pulmonary aspergillosis.

ELIGIBILITY:
Inclusion Criteria:

* 65ys≥age≥18ys
* renal transplant recipients

Exclusion Criteria:

* subjects with hypersensitivity to amphotericin B
* receipt of inhalational or intravenous amphotericin B within last 30 days
* subjects with known invasive fungal infection before renal transplant
* subjects with pneumonia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-09 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
invasive pulmonary aspergillosis | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital,Affiliate of Capital Medical University, Beijing, Beijing Municipality, China